CLINICAL TRIAL: NCT01695044
Title: A Phase 2, Open-label, Multicenter Study of PSMA ADC in Subjects With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of PSMA ADC in Subjects With Metastatic Castration-resistant Prostate Cancer (mCRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSMA ADC 2301
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PSMA ADC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: PSMA ADC (Experimental): Prostate Specific Membrane Antigen Antibody Drug Conjugate (PSMA ADC) administered IV at 2.5 mg/kg Q3W for 8 cycles or 2.3 mg/kg Q3W for 8 cycles.
  Interventions: Drug: PSMA ADC

INTERVENTIONS:
Drug: PSMA ADC — PSMA ADC administered IV at 2.5 mg/kg Q3W for 8 cycles or 2.3 mg/kg Q3W for 8 cycles.

SUMMARY:
PSMA ADC 2301 is a Phase 2, open-label, study to assess the anti-tumor activity and tolerability of Prostate Specific Membrane Antigen Antibody Drug Conjugate (PSMA ADC) in two groups of subjects with metastatic castration-resistant prostate cancer (mCRPC). One group comprises subjects who must have received at least one taxane-containing chemotherapy regimen (e.g. docetaxel, cabazitaxel). The second group comprises subjects who are cytotoxic chemotherapy-naïve. Subjects who are cytotoxic chemotherapy-naïve must have received and progressed on-, be ineligible for, refused, have an intolerance to-, or not have access to Radium-223. Both groups of subjects must also have received and progressed on abiraterone acetate and/or enzalutamide. If a subject is unable to receive abiraterone acetate and/or enzalutamide, Sponsor approval is required for participation in the study. Subjects will receive up to eight doses of PSMA ADC approximately once every three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of metastatic castration-resistant prostate cancer.
2. a) Prior history of treatment with at least one taxane-containing chemotherapy regimen (e.g. docetaxel, cabazitaxel). If a subject has received more than two cytotoxic chemotherapy regimens, Sponsor approval is required for study participation.

   OR

   b) No prior history of treatment with a cytotoxic chemotherapy regimen.
3. Must have received and progressed on abiraterone acetate and/or enzalutamide. If subject is unable to receive abiraterone acetate and/or enzalutamide, Sponsor approval is required for participation in the study.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
5. Life expectancy ≥ six months.
6. Cytotoxic chemotherapy-naïve subjects ONLY must have received and progressed on-, be ineligible for, refused, have an intolerance to-, or not have access to Radium-223.

Exclusion Criteria:

1. Treatment within 30 days prior to first dose of study drug of the following:

   * External Radiation therapy
   * Radiopharmaceuticals
   * Cytotoxic chemotherapy
   * Treatment with an investigational agent
2. Clinically significant cardiac disease or severe debilitating pulmonary disease
3. An acute infection requiring ongoing antibiotic therapy
4. Any prior treatment with PSMA ADC or other therapies targeting PSMA, or other antibody drug conjugate (ADC) products that contain monomethyl auristatin E (MMAE) (e.g., brentuximab vedotin, glembatumumab vedotin, ASG-5ME, RG7450) unless approved by Sponsor.
5. History of drug and/or alcohol abuse
6. History of pancreatitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Wong, PhD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (35):
- United States (35):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Burbank, California
  - Encinitas, California
  - Los Angeles, California
  - San Diego, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Norwalk, Connecticut
  - Port Saint Lucie, Florida
  - Honolulu, Hawaii
  - Fairway, Kansas
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lake Success, New York
  - New York, New York
  - Rochester, New York
  - Stony Brook, New York
  - Huntersville, North Carolina
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - Norfolk, Virginia
  - Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: PSMA ADC: PSMA ADC administered IV at 2.5 mg/kg Q3W for 8 cycles or 2.3 mg/kg Q3W for 8 cycles.
Period: Overall Study
Arm/Group | Arm 1: PSMA ADC
Started | 119
Completed | 17
Not Completed | 102

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: PSMA ADC Chemotherapy-experienced: PSMA ADC administered IV at 2.5 mg/kg Q3W for 8 cycles or 2.3 mg/kg Q3W for 8 cycles.
- Arm 2: PSMA ADC Chemotherapy-naive: PSMA ADC administered IV at 2.3 mg/kg Q3W for 8 cycles.
- Total: Total of all reporting groups
Arm/Group | Arm 1: PSMA ADC Chemotherapy-experienced | Arm 2: PSMA ADC Chemotherapy-naive | Total
Number analyzed (Participants) | 84 | 35 | 119
Age, Continuous [Mean (Full Range); unit: years] | 70.7 [50 to 91] | 73.1 [50 to 87] | 71.4 [50 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 84 | 35 | 119
Prostate specific antigen (PSA) [Mean (Standard Deviation); unit: ug/mL] | 804.8 (2173.38) | 220.9 (438.35) | 633.1 (1857.2)
PSA [Median (Full Range); unit: ug/mL] | 188.9 [7.5 to 17459.6] | 94.1 [1.4 to 2307.8] | 162.9 [1.4 to 17459.6]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Total Serum PSA Response
Description: Total serum prostate-specific antigen (PSA) response was defined as any decrease from baseline of at least 30% or 50%.
Time Frame: 24 Weeks
Population: Both groups must also have received and progressed on abiraterone acetate and/or enzalutamide prior to the study (once these agents were commercially available for use). The population examined was those subjects with a PSA baseline value and at least one post-baseline value.
Measure: Number; unit: % of responders
Groups:
- PSMA ADC Chemotherapy-experienced: Prostate Specific Membrane Antigen Antibody Drug Conjugate (PSMA ADC) administered IV at 2.3 mg/kg Q3W for 8 cycles.
  The chemotherapy-experienced group was comprised of 84 subjects who must have received at least one taxane-containing chemotherapy regimen (e.g., docetaxel, cabazitaxel) prior to the study (more than two cytotoxic chemotherapy regimens required sponsor approval for study participation).
- Chemotherapy-naive: Prostate Specific Membrane Antigen Antibody Drug Conjugate (PSMA ADC) administered IV at 2.3 mg/kg Q3W for 8 cycles.
  The chemotherapy-naïve group was comprised of 35 subjects who were cytotoxic chemotherapy-naïve. Chemotherapy-naïve subjects must have received and progressed on Radium-223 (following its approval by FDA), or have been ineligible for it, refused it, had an intolerance to it, or did not have access to it.
Arm/Group | PSMA ADC Chemotherapy-experienced | Chemotherapy-naive
Number analyzed (Participants) | 79 | 34
% of responders
  >30% Decrease in PSA | 29 | 32
  >50% Decrease in PSA | 11 | 21

2. Primary Outcome: CTC Response
Description: Circulating tumor cells (CTC) response was examined at two levels: at least 30% decrease or at least 50% decrease in CTC levels. Response was defined as any decrease from baseline of at least 30% or 50%.
Time Frame: 24 Weeks
Population: Both groups must also have received and progressed on abiraterone acetate and/or enzalutamide prior to the study (once these agents were commercially available for use). The population examined was those subjects with a CTC baseline value and at least one post-baseline value.
Measure: Number; unit: % of responders
Groups:
- PSMA ADC Chemotherapy-experienced: PSMA ADC administered IV at 2.3 mg/kg Q3W for 8 cycles.
  The chemotherapy-experienced group was comprised of 84 subjects who must have received at least one taxane-containing chemotherapy regimen (e.g., docetaxel, cabazitaxel) prior to the study (more than two cytotoxic chemotherapy regimens required sponsor approval for study participation).
- Chemotherapy-naive: PSMA ADC administered IV at 2.3 mg/kg Q3W for 8 cycles.
  The chemotherapy-naïve group was comprised of 35 subjects who were cytotoxic chemotherapy-naïve. Chemotherapy-naïve subjects must have received and progressed on Radium-223 (following its approval by FDA), or have been ineligible for it, refused it, had an intolerance to it, or did not have access to it.
Arm/Group | PSMA ADC Chemotherapy-experienced | Chemotherapy-naive
Number analyzed (Participants) | 68 | 26
% of responders
  >30% Decrease in CTC | 81 | 92
  >50% Decrease in CTC | 74 | 85

3. Primary Outcome: Overall Radiologic Response
Description: Overall radiologic response was measured prior to the first dose of study drug, at predose of cycle 5, and at the end of study. Imaging techniques used at screening were used throughout the study. The preferred imaging techniques include: bone scan, contrast enhanced CT of chest, contrast enhanced CT of pelvis, and contrast enhanced CT of upper & lower abdomen. Best overall radiologic response (confirmed), target and non-target lesions, was defined as responses in bone, visceral or nodal metastases according to the Modified Response Evaluation Criteria (RECIST 1.1). The best overall radiologic response is the best response recorded from the start of the treatment until disease progression/recurrence (taking, as reference for progressive disease, the smallest measurements recorded since the treatment started). The subject's best response assignment depended on the achievement of both measurement and confirmation criteria.
Time Frame: 24 weeks
Population: Both groups must also have received and progressed on abiraterone acetate and/or enzalutamide prior to the study (once these agents were commercially available for use). The full modified Intention-to-Treat (mITT) population (n = 119) was examined.
Measure: Number; unit: % of subjects
Arm/Group | PSMA ADC Chemotherapy-experienced | Chemotherapy-naive
Number analyzed (Participants) | 84 | 35
% of subjects
  Non-evaluable | 26 | 17
  Partial response | 0 | 6
  Progressive disease | 13 | 9
  Stable disease | 61 | 69

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | PSMA ADC Chemotherapy-experienced | Chemotherapy-naive
Serious Adverse Events (participants affected / at risk) | 43/84 | 18/35
Other Adverse Events (participants affected / at risk) | 84/84 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PSMA ADC Chemotherapy-experienced (N=84) | Chemotherapy-naive (N=35)
Anemia (Blood and lymphatic system disorders) | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Hemorrhagic anemia (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Ileus (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 3 | 0
Fatigue (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Bacteremia (Infections and infestations) | 2 | 0
Lobar pneumonia (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 2 | 1
ECG QT prolonged (Investigations) | 2 | 0
Decreased neutrophil count (Investigations) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 5
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 1 | 2
Acute renal failure (Renal and urinary disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PSMA ADC Chemotherapy-experienced (N=84) | Chemotherapy-naive (N=35)
Anemia (Blood and lymphatic system disorders) | 25 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 16 | 6
Tachycardia (Cardiac disorders) | 2 | 2
Vertigo (Cardiac disorders) | 3 | 2
Vision blurred (Eye disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 41 | 23
Diarrhea (Gastrointestinal disorders) | 33 | 16
Constipation (Gastrointestinal disorders) | 30 | 12
Vomiting (Gastrointestinal disorders) | 22 | 12
Abdominal pain (Gastrointestinal disorders) | 15 | 5
Dyspepsia (Gastrointestinal disorders) | 7 | 6
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 2
Flatulence (Gastrointestinal disorders) | 4 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 | 1
Fatigue (General disorders) | 52 | 19
Peripheral edema (General disorders) | 18 | 4
Asthenia (General disorders) | 13 | 3
Pain (General disorders) | 9 | 3
Chills (General disorders) | 4 | 2
Gait disturbance (General disorders) | 5 | 2
Pyrexia (General disorders) | 6 | 2
Urinary tract infection (Infections and infestations) | 9 | 4
Upper resiratory tract infection (Infections and infestations) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 7 | 7
Excoriation (Injury, poisoning and procedural complications) | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 1
Aspartate aminotransferase increased (Investigations) | 18 | 1
Decreased neutrophil count (Investigations) | 14 | 3
Decreased weight (Investigations) | 14 | 8
Alanine aminotransferase increased (Investigations) | 10 | 1
White blood cell count decreased (Investigations) | 10 | 0
Blood alkaline phosphatase increased (Investigations) | 8 | 1
Lymphocyte count decreased (Investigations) | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 40 | 15
Dehydration (Metabolism and nutrition disorders) | 20 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 15 | 2
Hypokalemia (Metabolism and nutrition disorders) | 14 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 13 | 2
Hyponatremia (Metabolism and nutrition disorders) | 13 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 19 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Peripheral neuropathy (Nervous system disorders) | 31 | 13
Headache (Nervous system disorders) | 17 | 3
Dizziness (Nervous system disorders) | 11 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 8
Dysgeusia (Nervous system disorders) | 5 | 6
Ataxia (Nervous system disorders) | 3 | 2
Paraesthesia (Nervous system disorders) | 5 | 1
Sciatica (Nervous system disorders) | 0 | 2
Transient ischemic attack (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 18 | 6
Depression (Psychiatric disorders) | 3 | 5
Anxiety (Psychiatric disorders) | 5 | 3
Confusional state (Psychiatric disorders) | 5 | 1
Hematuria (Renal and urinary disorders) | 4 | 2
Proteinuria (Renal and urinary disorders) | 5 | 0
Acute renal failure (Renal and urinary disorders) | 1 | 3
Urinary incontinence (Renal and urinary disorders) | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 5
Rash (Skin and subcutaneous tissue disorders) | 4 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Deep vein thrombosis (Vascular disorders) | 3 | 2
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No